CLINICAL TRIAL: NCT03912259
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Dupilumab in Chinese Adult Patients With Moderate-to-severe Atopic Dermatitis
Brief Title: Evaluation of Dupilumab in Chinese Adult Patients With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC15116; U1111-1190-7728 (Other: UTN)
Record Dates: First submitted 2018-12-18; First posted 2019-04-11 (Actual); Results first posted 2021-04-05 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab; Emollients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo Q2W (Placebo Comparator): Placebo matched to dupilumab 600 milligrams (mg) (loading dose), subcutaneously (SC) on Day 1 followed by placebo matched to dupilumab 300 mg once every 2 weeks (Q2W) for 16 weeks.
  Interventions: Drug: Placebo; Drug: Emollient (moisturizer)
- Dupilumab 300 mg Q2W (Experimental): Dupilumab at a loading dose of 600 mg, SC on Day 1 followed by 300 mg, Q2W for 16 weeks.
  Interventions: Drug: Dupilumab; Drug: Emollient (moisturizer)

INTERVENTIONS:
Drug: Dupilumab — Pharmaceutical form: solution,
  Route of administration: SC
  Other Names: Dupixent; SAR231893
  Arms: Dupilumab 300 mg Q2W
Drug: Placebo — Pharmaceutical form: solution,
  Route of administration: SC
  Arms: Placebo Q2W
Drug: Emollient (moisturizer) — Pharmaceutical form: cream,
  Route of administration: topical use

SUMMARY:
Primary Objective:

To evaluate the efficacy of dupilumab monotherapy compared to placebo treatment in adult participants with moderate-to-severe atopic dermatitis (AD).

Secondary Objectives:

* To evaluate the safety of dupilumab monotherapy compared to placebo treatment in adult participants with moderate-to-severe AD.
* To evaluate the effect of dupilumab on improving patient reported outcomes (PROs).
* To evaluate dupilumab immunogenicity.

DETAILED DESCRIPTION:
The maximum study duration was 33 weeks per participants, including a screening period of up to 5 weeks, a 16-week randomized treatment period, and a 12-week follow-up period.

ELIGIBILITY:
Inclusion criteria:

* Male or female, 18 years or older.
* AD (according to American Academy of Dermatology Consensus Criteria, 2014) that had been present for at least 3 years before the screening visit.
* Eczema Area and Severity Index (EASI) score greater than or equal to (>=) 16 at the screening and baseline visits.
* Investigator's Global Assessment (IGA) score >=3 (on the 0 to 4 IGA scale, in which 3 was moderate and 4 was severe) at the screening and baseline visits.
* Participants with >=10 percent (%) body surface area (BSA) of AD involvement at the screening and baseline visits.
* Baseline Pruritus Numerical Rating Scale (NRS) average score for maximum itch intensity >=4.
* Documented recent history (within 6 months before the screening visit) of inadequate response to treatment with topical medications or for whom topical treatments were otherwise medically inadvisable (e.g., because of important side effects or safety risks).

Exclusion criteria:

* Had used any of the following treatments within 4 weeks before the baseline visit, or any condition that, in the opinion of the investigator, was likely to require such treatment(s) during the first 4 weeks of study treatment:

  * Immunosuppressive/immunomodulating drugs (e.g., systemic corticosteroids, cyclosporine, mycophenolate-mofetil, interferon-gamma [IFN-γ], Janus kinase inhibitors, azathioprine, methotrexate);
  * Phototherapy for AD.
* Treatment with topical corticosteroids (TCS) or topical calcineurin inhibitors (TCI) within 1 week before the baseline visit.
* Treatment with systemic Traditional Chinese Medicine (TCM) within 4 weeks before the baseline visit or treatment with topical TCM within 1 week before the baseline visit.
* Treatment with biologics as follows:

  * Any cell-depleting agents including but not limited to rituximab: within 6 months before the baseline visit, or until lymphocyte count returns to normal, whichever is longer;
  * Other biologics: within 5 half-lives (if known) or 16 weeks prior to baseline visit, whichever was longer.
* Initiation of treatment of AD with prescription moisturizers or moisturizers containing additives such as ceramide, hyaluronic acid, urea, or filaggrin degradation products during the screening period (participants may continue using stable doses of such moisturizers if initiated before the screening visit).
* Regular use (more than 2 visits per week) of a tanning booth/parlor within 4 weeks of the baseline visit.
* Treatment with a live (attenuated) vaccine within 12 weeks before the baseline visit.
* Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 2 weeks before the baseline visit, or superficial skin infections within 1 week before the baseline visit. NOTE: participants may be rescreened after infection resolves.
* Known or suspected history of immunosuppression, including history of invasive opportunistic infections (e.g., tuberculosis [TB], histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis) despite infection resolution: or unusually frequent, recurrent, or prolonged infections, per investigator judgment.
* Active TB, latent untreated TB or a history of incompletely treated TB or non-tuberculous mycobacterial infection were excluded from the study unless that was well documented by a specialist that the participants had adequately treated and could then start treatment with a biologic agent, in the medical judgment of the Investigator and/or infectious disease specialist. TB testing would be performed according to local guidelines if required by regulatory authorities or ethics committees.

The above information was not intended to contain all considerations relevant to a participants potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (27):
- China (27):
  - Investigational Site Number 1560019, Beijing
  - Investigational Site Number 1560001, Beijing
  - Investigational Site Number 1560004, Beijing
  - Investigational Site Number 1560003, Beijing
  - Investigational Site Number 1560010, Beijing
  - Investigational Site Number 1560021, Changchun
  - Investigational Site Number 1560006, Changsha
  - Investigational Site Number 1560017, Chongqing
  - Investigational Site Number 1560026, Hangzhou
  - Investigational Site Number 1560007, Hangzhou
  - Investigational Site Number 1560013, Jinan
  - Investigational Site Number 1560020, Kunming
  - Investigational Site Number 1560030, Lianyungang
  - Investigational Site Number 1560022, Nanjing
  - Investigational Site Number 1560029, Ningbo
  - Investigational Site Number 1560016, Shanghai
  - Investigational Site Number 1560023, Shanghai
  - Investigational Site Number 1560018, Shanghai
  - Investigational Site Number 1560015, Shanghai
  - Investigational Site Number 1560002, Shenyang
  - Investigational Site Number 1560005, Shenyang
  - Investigational Site Number 1560008, Shenyang
  - Investigational Site Number 1560024, Shenzhen
  - Investigational Site Number 1560027, Tianjin
  - Investigational Site Number 1560028, Wuxi
  - Investigational Site Number 1560012, Xi'an
  - Investigational Site Number 1560025, Yancheng

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Mickevicius T, Pink AE, Bhogal M, O'Brart D, Robbie SJ. Dupilumab-Induced, Tralokinumab-Induced, and Belantamab Mafodotin-Induced Adverse Ocular Events-Incidence, Etiology, and Management. Cornea. 2023 Apr 1;42(4):507-519. doi: 10.1097/ICO.0000000000003162. Epub 2022 Dec 15. PMID 36525340

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 25 active centers in China between 19 Dec 2018 and 14 Feb 2020. A total of 165 participants were randomized and treated in the study.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to dupilumab or placebo according to a central randomization scheme provided by an interactive response technology.
Period: Overall Study
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Started | 83 | 82
Completed | 66 | 76
Not Completed | 17 | 6
Not completed — Adverse Event (AE) | 2 | 4
Not completed — Lack of Efficacy | 4 | 1
Not completed — Withdrawal by Subject | 11 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Intent-to-treat (ITT) population which consisted of all randomized participants.
Groups:
- Placebo Q2W: Placebo matched to dupilumab 600 mg (loading dose), SC on Day 1 followed by placebo matched to dupilumab 300 mg Q2W for 16 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W | Total
Number analyzed (Participants) | 83 | 82 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (12.46) | 31.0 (10.47) | 30.6 (11.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 60 | 58 | 118
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 83 | 82 | 165
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Investigator's Global Assessment (IGA) Score [Count of Participants; unit: Participants] — The IGA is an assessment instrument used to rate the severity of atopic dermatitis (AD) globally based on a 5-point scale ranging from (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe), where higher score indicated higher severity.
  Participants
    IGA = 3 | 37 | 35 | 72
    IGA = 4 | 46 | 47 | 93

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Investigator's Global Assessment (IGA) Score of "0" or "1" and Reduction From Baseline of Greater Than or Equal to (>=) 2 Points at Week 16
Description: The IGA is an assessment instrument used to rate the severity of AD globally based on a 5-point scale ranging from (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe), higher score indicated higher severity.
Time Frame: Baseline, Week 16
Population: Analysis was performed on ITT population.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Q2W: Placebo matched to dupilumab 600 mg (loading dose), SC on Day 1 followed by placebo matched to dupilumab 300 mg, Q2W for 16 weeks.
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
Participants | 4 | 22
Statistical Analysis 1: Comparison: Placebo Q2W vs Dupilumab 300 mg Q2W; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; P-value was derived by the Cochran-Mantel-Haenszel test stratified by baseline disease severity (IGA=3 vs. IGA=4); Difference in Percentage = 22.0, 95% CI 2-sided [11.37 to 32.65]

2. Secondary Outcome: Number of Participants With Eczema Area and Severity Index (EASI) - 75 Response (>= 75% Reduction in Score From Baseline) at Week 16
Description: EASI: Measure to assess severity and extent of AD based on 4 AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation] and lichenification). Each characteristic was assessed for severity by Investigator/designee on scale of "0" (absent) through "3" (severe) and scored separately for each of 4 body regions (head, trunk, upper and lower extremities). Total score range from 0 (minimum) to 72 (maximum), higher scores indicated greater severity of AD.
Time Frame: Baseline, Week 16
Population: Analysis was performed on ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
Participants | 12 | 47

3. Secondary Outcome: Number of Participants Who Achieved >=4 Points With Reduction From Baseline in Weekly Average of Peak Daily Pruritus Numerical Rating Scale (NRS) Score at Week 16
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]), higher scores indicated greater severity.
Time Frame: Baseline, Week 16
Population: Analysis was performed on ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
Participants | 4 | 32

4. Secondary Outcome: Number of Participants Who Achieved >=3 Points With Reduction From Baseline in Weekly Average of Peak Daily Pruritus Numerical Rating Scale Score at Week 16
Description: as for outcome 3
Time Frame: Baseline, Week 16
Population: Analysis was performed on ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
Participants | 8 | 43

5. Secondary Outcome: Percentage Change From Baseline at Week 16 in Weekly Average of Peak Daily Pruritus NRS
Description: as for outcome 3
Time Frame: Baseline, Week 16
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
percentage change | -21.13 (3.610) | -48.59 (3.026)

6. Secondary Outcome: Change From Baseline at Week 16 in Weekly Average of Peak Daily Pruritus NRS
Description: as for outcome 3
Time Frame: Baseline, Week 16
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
units on a scale | -1.64 (0.272) | -3.84 (0.237)

7. Secondary Outcome: Percentage Change From Baseline to Week 16 in EASI Score
Description: EASI: Measure to assess severity & extent of AD based on 4 AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation] & lichenification). Each characteristic was assessed for severity by Investigator/designee on scale of "0" (absent) through "3"(severe) & scored separately for each of 4 body regions (head, trunk, upper & lower extremities). Total score ranges from 0 (minimum) to 72 (maximum), higher scores indicated greater severity of AD.
Time Frame: Baseline to Week 16
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
percentage change | -39.44 (4.936) | -75.23 (3.879)

8. Secondary Outcome: Change From Baseline to Week 16 in Percent Body Surface Area (BSA) of AD Involvement
Description: BSA affected by AD was assessed for each section of the body (the possible highest score for each region was: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]) and reported as a percentage of all major body sections combined. The reported percentage of BSA was combined percentage of all major body sections.
Time Frame: Baseline to Week 16
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: percentage of body surface area
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
percentage of body surface area | -19.25 (2.557) | -37.76 (2.126)

9. Secondary Outcome: Change From Baseline to Week 16 in Dermatology Life Quality Index (DLQI) Total Score
Description: The DLQI was a validated questionnaire used to measure the impact of AD disease symptoms and treatment on health-related quality of life (QOL). DLQI consisting of a set of 10 questions which assess QOL over the past week. Responses to each questions were assessed on a scale of 0 to 3, where 0 is "not at all" and 3 is "very much". Scores from all 10 questions added up to give total DLQI scores ranged from 0 (not at all) to 30 (very much), higher scores indicated more impact on quality of life.
Time Frame: Baseline to Week 16
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
units on a scale | -5.06 (0.701) | -10.33 (0.625)

10. Secondary Outcome: Change From Baseline to Week 16 in Patient Oriented Eczema Measure (POEM)
Description: The POEM is a 7-item self-assessment questionnaire that assesses disease symptoms on a scale ranging from 0 to 4 (0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, 4 = all days). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (severe disease). Higher scores indicated more severe disease and poor quality of life.
Time Frame: Baseline to Week 16
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
units on a scale | -4.04 (0.788) | -12.89 (0.685)

11. Secondary Outcome: Percentage Change From Baseline to Week 2 in Weekly Average of Peak Daily Pruritus NRS
Description: as for outcome 3
Time Frame: Baseline to Week 2
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
percentage change | -4.75 (1.802) | -15.65 (1.818)

12. Secondary Outcome: Percentage Change From Baseline to Week 16 in EuroQoL Five Dimensions Questionnaire (EQ-5D) Index Scores
Description: The EQ-5D is a standardized measure of health status which is consists of 2 parts; the descriptive system and the EQ visual analogue scale (EQVAS). The EQ-5D descriptive system includes 5 dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension measured on 3 levels: "no problem" (level 1), "some problems" (level 2), "extreme problems" (level 3). The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state. The 5 dimensional 3-level systems was converted into single index utility score between 0 to 1 that quantify health status, where 0 represents "death" and 1 represents "perfect health".
Time Frame: Baseline to Week 16
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
percentage change | 2.92 (0.692) | 8.00 (0.562)

13. Secondary Outcome: Percentage Change From Baseline to Week 16 in EuroQoL Five Dimensions Questionnaire Visual Analog Scale Scores
Description: The EQ-5D VAS records the respondent's self-rated health on a vertical, visual analogue scale ranged from 0-100 where 100 indicated "best imaginable health state" and 0 indicated "worst imaginable health state", higher scores indicated better outcome.
Time Frame: Baseline to Week 16
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
percentage change | 60.19 (25.154) | 90.32 (24.775)

14. Secondary Outcome: Absolute Change From Baseline to Week 16 in EQ-5D Index Scores
Description: The EQ-5D is a standardized measure of health status which consisted of 2 parts; the descriptive system and the EQVAS. The EQ-5D descriptive system includes 5 dimensions; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension measured on 3 levels: "no problem" (level 1), "some problems" (level 2), "extreme problems" (level 3). The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state. The 5 dimensional 3-level systems was converted into single index utility score between 0 to 1 that quantify health status, where 0 represents "death" and 1 represents "perfect health".
Time Frame: Baseline to Week 16
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
units on a scale | 0.02 (0.006) | 0.06 (0.004)

15. Secondary Outcome: Absolute Change From Baseline to Week 16 in EuroQoL Five Dimensions Questionnaire Visual Analog Scale Scores
Description: as for outcome 13
Time Frame: Baseline to Week 16
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
units on a scale | 10.75 (2.689) | 18.22 (2.243)

16. Secondary Outcome: Number of Participants Who Achieve Reduction of IGA Score by >=2 From Baseline to Week 16
Description: The IGA is an assessment instrument used to rate the severity of AD globally, based on a 5-point scale ranging from (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe), higher score indicated higher severity. In this outcome measure, number of participants who achieved reduction from baseline of >=2 points in IGA score at Week 16 were reported.
Time Frame: Baseline to Week 16
Population: Analysis was performed on ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
Participants | 7 | 39

17. Secondary Outcome: Number of Participants Achieving IGA 0 to 1 and a Reduction of >=2 Points From Baseline Through Week 16
Description: as for outcome 1
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
Population: Analysis was performed on ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
Participants
  Week 2 | 0 | 2
  Week 4 | 0 | 6
  Week 8 | 0 | 9
  Week 12 | 4 | 16
  Week 16 | 4 | 22

18. Secondary Outcome: Absolute Change in EASI Score From Baseline at Weeks 2, 4, 8, 12 and 16
Description: EASI: Measure to assess severity & extent of AD based on 4 AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation] & lichenification). Each characteristic was assessed for severity by Investigator/designee on scale of "0" (absent) through "3" (severe) & scored separately for each of 4 body regions (head, trunk, upper & lower extremities). Total score range from 0 (minimum) to 72 (maximum), higher scores indicated greater severity of AD. Participants with missing EASI Score at each visit were imputed using MI (Multiple Imputation) method.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
Population: Analysis was performed on ITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
units on a scale
  Week 2 | -3.27 (7.974) | -12.48 (12.640)
  Week 4 | -6.45 (11.838) | -19.56 (13.687)
  Week 8 | -9.54 (10.947) | -22.45 (12.830)
  Week 12 | -11.23 (12.603) | -24.32 (14.191)
  Week 16 | -12.60 (12.484) | -25.87 (13.985)

19. Secondary Outcome: Percentage Change in EASI Score From Baseline at Weeks 2, 4, 8, 12 and 16
Description: EASI: Measure to assess severity & extent of AD based on 4 AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation] & lichenification). Each characteristic was assessed for severity by Investigator/designee on scale of "0" (absent) through "3" (severe) & scored separately for each of 4 body regions (head, trunk, upper & lower extremities). Total score range from 0 (minimum) to 72 (maximum), higher scores indicated greater severity of AD.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12, Week 16
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
percentage change
  Week 2 | -10.55 (2.977) | -35.69 (2.930)
  Week 4 | -19.28 (3.981) | -55.83 (3.684)
  Week 8 | -29.38 (4.147) | -65.84 (3.562)
  Week 12 | -35.26 (4.674) | -70.36 (4.047)
  Week 16 | -39.44 (4.936) | -75.23 (3.879)

20. Secondary Outcome: Number of Participants With EASI-50 (>=50% Improvement From Baseline) at Week 16
Description: as for outcome 19
Time Frame: Baseline, Week 16
Population: Analysis was performed on ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
Participants | 24 | 58

21. Secondary Outcome: Number of Participants With EASI-90 (>=90% Improvement From Baseline) at Week 16
Description: as for outcome 19
Time Frame: Baseline, Week 16
Population: Analysis was performed on ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
Participants | 5 | 33

22. Secondary Outcome: Absolute Change in Weekly Average of Peak Daily Pruritus NRS Score From Baseline Through Week 16
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]), higher scores indicated greater severity. Participants with missing Peak Daily Pruritus NRS Score at each visit were imputed using MI method.
Time Frame: From Baseline Through Week 16
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
units on a scale
  Week 1 | -0.26 (0.106) | -0.63 (0.107)
  Week 2 | -0.38 (0.135) | -1.26 (0.136)
  Week 3 | -0.61 (0.153) | -1.90 (0.153)
  Week 4 | -0.69 (0.162) | -2.26 (0.159)
  Week 5 | -0.88 (0.191) | -2.61 (0.187)
  Week 6 | -0.96 (0.205) | -2.81 (0.201)
  Week 7 | -0.88 (0.214) | -3.14 (0.208)
  Week 8 | -1.04 (0.212) | -3.21 (0.205)
  Week 9 | -1.10 (0.218) | -3.29 (0.209)
  Week 10 | -1.12 (0.221) | -3.38 (0.210)
  Week 11 | -1.24 (0.231) | -3.52 (0.216)
  Week 12 | -1.34 (0.233) | -3.59 (0.213)
  Week 13 | -1.46 (0.246) | -3.65 (0.223)
  Week 14 | -1.53 (0.264) | -3.71 (0.241)
  Week 15 | -1.56 (0.262) | -3.81 (0.234)
  Week 16 | -1.64 (0.272) | -3.84 (0.237)

23. Secondary Outcome: Percentage Change in Weekly Average of Peak Daily Pruritus NRS Score From Baseline Through Week 16
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]), higher scores indicated greater severity. Participants with missing peak NRS scores at each visit were imputed using MI method.
Time Frame: From Baseline Through Week 16
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
percentage change
  Week 1 | -2.95 (1.387) | -7.30 (1.405)
  Week 2 | -4.75 (1.802) | -15.65 (1.818)
  Week 3 | -7.92 (2.000) | -23.66 (1.988)
  Week 4 | -9.10 (2.118) | -28.17 (2.069)
  Week 5 | -11.56 (2.477) | -32.65 (2.410)
  Week 6 | -12.41 (2.623) | -35.01 (2.543)
  Week 7 | -11.37 (2.743) | -39.16 (2.642)
  Week 8 | -13.22 (2.710) | -40.36 (2.594)
  Week 9 | -14.03 (2.796) | -41.28 (2.655)
  Week 10 | -14.24 (2.857) | -42.51 (2.682)
  Week 11 | -15.72 (2.972) | -44.26 (2.746)
  Week 12 | -17.07 (3.048) | -45.37 (2.735)
  Week 13 | -18.80 (3.235) | -46.15 (2.845)
  Week 14 | -19.63 (3.501) | -47.04 (3.061)
  Week 15 | -19.96 (3.503) | -48.29 (3.009)
  Week 16 | -21.13 (3.610) | -48.59 (3.026)

24. Secondary Outcome: Number of Participants Who Responded "Absence of Pruritus" or "Mild Pruritus" in the Pruritus Categorical Scale at Week 16
Description: The pruritus categorical scale was a 4-point scale used to assess symptoms of AD. The scale is rated as follows: 0: absence of pruritus; 1: mild pruritus (occasional slight itching/scratching); 2: moderate pruritus (constant or intermittent itching/scratching that does not disturb sleep) and 3: severe pruritus (bothersome itching/scratching that disturbs sleep), higher scores indicated worse outcome.
Time Frame: Week 16
Population: Analysis was performed on ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 83 | 82
Participants | 12 | 49

25. Secondary Outcome: Number of Days of Sick Leave/Missed School Days
Description: Participants who were employed or enrolled in school for full time were asked to report the number of sick leave/missed school days since the last study assessment. Participants were counted as Full time if the participant checked "Full time" at all visits through 16-week treatment period and participants were counted as Part time if the participant checked at least one "Part time" during 16-week treatment period.
Time Frame: Week 16
Population: Analysis was performed on ITT population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' represent the number of participants analyzed for each specified row.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 58 | 66
Days
  Full time: number analyzed (Participants) | 47 | 58
  Full time | 0.66 (2.075) | 0.88 (3.468)
  Part time: number analyzed (Participants) | 11 | 8
  Part time | 11.14 (20.923) | 7.44 (9.202)

26. Secondary Outcome: Percentage of Participants With at Least One Day Sick Leave/Missed School Days
Description: as for outcome 25
Time Frame: Week 16
Population: as for outcome 25
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
Number analyzed (Participants) | 58 | 66
percentage of participants
  Full time: number analyzed (Participants) | 47 | 58
  Full time | 14.9 | 22.4
  Part time: number analyzed (Participants) | 11 | 8
  Part time | 72.7 | 75.0

ADVERSE EVENTS:
Time Frame: All AEs were collected from signature of the informed consent form up to end of study regardless of seriousness or relationship to investigational product. Time frame for reporting of treatment emergent adverse events (TEAEs) was from first dose up to 28 weeks.
Description: TEAEs are defined as AEs that developed or worsened during the treatment-emergent period. Safety population included all randomized participants received any investigational medicinal product (IMP). Participants were analyzed according to the treatment they actually received (as treated).
Arm/Group | Placebo Q2W | Dupilumab 300 mg Q2W
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/82
Serious Adverse Events (participants affected / at risk) | 4/83 | 1/82
Other Adverse Events (participants affected / at risk) | 57/83 | 56/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Q2W (N=83) | Dupilumab 300 mg Q2W (N=82)
Anaphylactic Reaction (Immune system disorders) | 1 (1) | 0 (0)
Connective Tissue Disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Q2W (N=83) | Dupilumab 300 mg Q2W (N=82)
Conjunctivitis Allergic (Eye disorders) | 1 (1) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 5 (5)
Conjunctivitis (Infections and infestations) | 4 (4) | 8 (8)
Folliculitis (Infections and infestations) | 6 (6) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 6 (8)
Upper Respiratory Tract Infection (Infections and infestations) | 10 (13) | 14 (16)
Blood Uric Acid Increased (Investigations) | 5 (6) | 1 (1)
Protein Urine Present (Investigations) | 9 (9) | 9 (10)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 41 (54) | 36 (51)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT03912259/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT03912259/SAP_001.pdf